CLINICAL TRIAL: NCT04289324
Title: Open Lung Maneuvers During High Frequency Oscillatory Ventilation in Extremely Preterm Infants - a Single Center Randomized Controlled Trial
Brief Title: Open Lung Maneuvers During High Frequency Oscillatory Ventilation in Preterm Infants
Acronym: OPEN4HFOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Tobias Werther, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1161/2019
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: High Frequency Oscillation Ventilation; Extreme Prematurity; Lung Injury, Acute
MeSH Terms: conditions — Acute Lung Injury

STUDY DESIGN:
Intervention Model Description: Single center randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): lung recruitment maneuvers performed every twelve hours during HFOV
  Interventions: Procedure: regular lung recruitment
- Control (No Intervention): no regular lung recruitment maneuvers during HFOV

INTERVENTIONS:
Procedure: regular lung recruitment — stepwise oxygenation-guided lung recruitment at regular (twelve hours) intervals during high frequency oscillation ventilation
  Arms: Intervention

SUMMARY:
To assess whether stepwise oxygenation-guided lung recruitment at regular intervals reduces the oxygen saturation index (OSI = Mean Airway Pressure × Fraction of inspired Oxygen × 100 / peripheral Oxygen Saturation, OSI = MAPxFiO2x100/SpO2) averaged over high frequency oscillation ventilation (HFOV) time in extremely preterm infants.

DETAILED DESCRIPTION:
Background: Open lung maneuvers aim to recruit and stabilize the majority of collapsed alveoli, using oxygenation as an indirect variable for lung volume. The stepwise oxygenation-guided lung recruitment procedure during frequency oscillatory ventilation (HFOV) in preterm infants has a low risk of lung hyperinflation and air leak syndrome. Nevertheless, open lung maneuvers at regular intervals during HFOV to maintain or restore oxygenation is not implemented as a routine procedure in the neonatal intensive care.

Aim of the study: To assess whether stepwise oxygenation-guided lung recruitment at regular intervals reduces the oxygen saturation index (OSI = Mean Airway Pressure × Fraction of inspired Oxygen × 100 / peripheral Oxygen Saturation, OSI = MAPxFiO2x100/SpO2) averaged over HFOV time in extremely preterm infants.

Study design: Single center randomized controlled study.

Methods: Thirty-six extremely preterm infants below 28 weeks of gestational age and on high frequency oscillation ventilation receive either stepwise oxygenation-guided lung recruitment maneuver at regular intervals (intervention) and upon decision of the care giving team (intervention group) or lung recruitment maneuver only upon decision of the care giving team (standard, control group). The primary outcome is the oxygen saturation index averaged over HFO ventilation time. The observation time of the HFOV will be limited to at most seven days.

Sample size: Fifteen infants need to be enrolled in each group to have 80% power (at a two-sided alpha level of 5%) to detect a difference of 25% in the oxygen saturation index between the intervention group and the control group.

Main outcome variables: Oxygen saturation index averaged over HFO ventilation time.

Secondary outcome variables: Bronchopulmonary dysplasia (BPD); days of ventilation; oxygen saturation index averaged over ventilation time (HFO and conventional ventilation); the following variables measured before, during and after a single stepwise oxygenation-guided recruitment maneuver: echocardiographic parameters, reactance, relative impedance changes, lung ultrasound measurements, transcutaneous partial carbon dioxide (CO2), blood pressure, heart rate.

ELIGIBILITY:
Inclusion Criteria: Preterm infants

* born below 28 weeks of gestational age
* not older than 29 weeks of postmenstrual age
* receive HFOV

Exclusion Criteria:

* known congenital anomalies of the heart, of the lung, and/or of the central nervous system
* known chromosomal abnormalities
* participation in other intervention trials

Max Age: 8 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HFOV oxygen saturation index | through study completion, an average 10 weeks
  oxygen saturation index averaged over high frequency oscillation ventilation for not more than seven consecutive days

SECONDARY OUTCOMES:
bronchopulmonary dysplasia | through study completion, an average 10 weeks
  respiratory support at 36 weeks postmenstrual age
days of ventilation | through study completion, an average 10 weeks
  days on conventional and high frequency oscillation ventilation
overall oxygen saturation index | through study completion, an average 10 weeks
  oxygen saturation index averaged over ventilation time

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Werther, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rimensberger PC, Pache JC, McKerlie C, Frndova H, Cox PN. Lung recruitment and lung volume maintenance: a strategy for improving oxygenation and preventing lung injury during both conventional mechanical ventilation and high-frequency oscillation. Intensive Care Med. 2000 Jun;26(6):745-55. doi: 10.1007/s001340051242. PMID 10945393
- [Background] Rimensberger PC, Beghetti M, Hanquinet S, Berner M. First intention high-frequency oscillation with early lung volume optimization improves pulmonary outcome in very low birth weight infants with respiratory distress syndrome. Pediatrics. 2000 Jun;105(6):1202-8. doi: 10.1542/peds.105.6.1202. PMID 10835058
- [Background] De Jaegere A, van Veenendaal MB, Michiels A, van Kaam AH. Lung recruitment using oxygenation during open lung high-frequency ventilation in preterm infants. Am J Respir Crit Care Med. 2006 Sep 15;174(6):639-45. doi: 10.1164/rccm.200603-351OC. Epub 2006 Jun 8. PMID 16763218
- [Background] de Waal K, Evans N, van der Lee J, van Kaam A. Effect of lung recruitment on pulmonary, systemic, and ductal blood flow in preterm infants. J Pediatr. 2009 May;154(5):651-5. doi: 10.1016/j.jpeds.2009.01.012. PMID 19364558
- [Background] Zannin E, Doni D, Ventura ML, Fedeli T, Rigotti C, Dellaca RL, Tagliabue PE. Relationship between Mean Airways Pressure, Lung Mechanics, and Right Ventricular Output during High-Frequency Oscillatory Ventilation in Infants. J Pediatr. 2017 Jan;180:110-115. doi: 10.1016/j.jpeds.2016.09.015. Epub 2016 Oct 10. PMID 27745747
- [Derived] Werther T, Kueng E, Aichhorn L, Pummer L, Goeral K, Berger A, Hermon M, Klebermass-Schrehof K. Regular lung recruitment maneuvers during high-frequency oscillatory ventilation in extremely preterm infants: a randomized controlled trial. BMC Pediatr. 2022 Dec 12;22(1):710. doi: 10.1186/s12887-022-03780-7. PMID 36503480